CLINICAL TRIAL: NCT04238377
Title: Evaluation of Post Mastectomy Pain Syndrome After Preoperative Stellate Ganglion Block for Breast Cancer Surgeries, Clinical Randomized Controlled Trial
Brief Title: Post Mastectomy Pain Syndrome After Preoperative Stellate Ganglion Block for Breast Cancer Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Ahmed Salman Solyman Salman, Aneasthetist, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201617048.3
Record Dates: First submitted 2020-01-19; First posted 2020-01-23 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Breast Cancer; Breast Pain
Keywords: Stellate Ganglion Block , Neuropathic pain syndromes
MeSH Terms: conditions — Breast Neoplasms; Mastodynia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stellate Group (Active Comparator): will receive pre-operative ultrasound guided stellate ganglion block one hour before surgery and multimodal analgesia and will be followed for 6 months for neuropathic pain as the Stellate Group
  Interventions: Procedure: Stellate Ganglion Block; Drug: Multimodal Analgesia
- Control Group (Placebo Comparator): will receive multimodal analgesia only and will be followed for 6 months for neuropathic pain as the control Group
  Interventions: Drug: Multimodal Analgesia

INTERVENTIONS:
Procedure: Stellate Ganglion Block — Using US with a linear array transduce, subfascial-C6- Stellate Ganglion Block. Patients will be supine with the neck slightly hyper- extended. After aseptic preparation of the skin, the transducer is placed on the neck to enable cross sectional visualization of anatomical structures at the level of C6. The carotid artery, internal jugular vein, thyroid gland, trachea, longus colli covered with the prevertebral fascia, root of C6, and transverse process of C6 are all visualized. The transducer will then gently be pressed between the carotid artery and trachea to retract the carotid artery laterally and to position the transducer close to the longus colli.
  A 1.0-inch, 25-gauge long-bevel needle were paratracheal inserted toward the middle of the longus colli. The endpoint for injection were the ultrasound image demonstrating the tip of needle penetrating the prevertebral fascia in the longus colli. After negative aspiration, 5 mL of 0.5% bupivacaine was injected
  Other Names: Cervicothoracic Ganglion Block
  Arms: Stellate Group
Drug: Multimodal Analgesia — Multimodal analgesia in the form of administering of IV paracetamol 1000 mg one hour prior to start of surgery in combination 30 mg ketorolac and Single preoperative 0.1 mg/kg dose dexamethasone has a combined action, anti-emetic and provides enhanced analgesia, with intra-operative fast acting opioid analgesics, Fentanyl 2 mic/kg
  Other Names: Preventive Analgesia

SUMMARY:
This study investigate the effect of pre-operative ultrasound guided stellate ganglion block with local anesthetic on the frequency of neuropathic pain syndromes in the first 6-month post cancer breast surgeries with axillary dissection.

DETAILED DESCRIPTION:
In this study Eighty Female patients with a diagnosis of breast cancer, underwent breast surgery with axillary dissection at National Cancer Institute, Cairo University were included in this study. Patients will be randomized into two equal comparable groups of patients.

(Group A the study group) was received pre-operative ultrasound guided stellate ganglion block one hour before surgery and multimodal analgesia and (Group B the control group) was received multimodal analgesia only.

The present study showed in regards to the acute pain management of the stellate ganglion block: intraoperative hemodynamics, mean arterial blood pressure and heart rate (MABP, HR) were statistically significant less in group A (Stellate Group) than group B (Control Group) and this leads to significant less opioid consumption in Group A (Stellate Group) than Group B (Control group). In the 1st 24h postoperative opioid consumption measured by number of rescue dose of morphine 5mg IV were administered when visual analogue score was more than 4 and total requirement per 24 hours was recorded. The results show statistically significant less opioid consumption in Group A (Stellate Group) with average visual analogue score 3.5 in 1st 24h than Group B (Control group) with average visual analogue score 5.5 in 1st 24h.

The present study showed in regards to the chronic pain management of the stellate ganglion block that, the 6-month relative frequency of neuropathic pain syndromes, using the grading system for neuropathic pain (GSNP) shows statistically significance lower frequency of neuropathic pain syndromes in Group A (Stellate Group) than Group B (Control group).

Assessment of patient daily activity and functional capacity using Eastern cooperative oncology group (ECOG) scoring showed statistically significance higher performance status (lower numbers in the score) in Group A (Stellate Group) than Group B (Control group).

Number of patients discharged on tramadol & or Lyrica whom developed Post Mastectomy Pain syndrome (PMPs) is statically significant lower in Group A (Stellate Group) than Group B (Control group).

ELIGIBILITY:
Inclusion Criteria:

* Women were eligible if a diagnosis of breast cancer, programmed for breast surgery with axillary dissection, able to understand and willing to follow the study protocol

Exclusion Criteria:

* Patient refusal - Local infection at the site of injection - Allergy to study medications - Psychosocial disorders - pts on opioid or antianxiety - Sepsis - Anatomic abnormalities - Systemic anticoagulation or coagulopathy - Inability to comprehend or participate in pain scoring system - Recent myocardial infarction - Pathological bradycardia - Glaucoma
* Any contraindication for the multimodal analgesia e.g. (asthmatic patient and use of diclofenac, Diabetic patient and use of steroids)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-12-26 (Actual); Primary Completion 2020-03-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Neuropathic pain Syndromes | 6 months after surgery
  relative frequency of neuropathic pain syndromes post breast surgeries with axillary dissection after preoperative ultrasound stellate ganglion block. This is accomplished using the grading system for neuropathic pain (GSNP),0: No Pain,1: Pain, 2: Possible neuropathic: Pain with (A history of relevant neurological lesion or disease AND Pain distribution neuroanatomically plausible, 3: Pain Probable neuropathic: Positive sensory signs (allodynia, hyperalgesia, electric, burning, numbness, itching, maybe motor or autonomic changes) on the distribution of the injured nerves or beyond, 4: Pain Definitive neuropathic: diagnostic test confirms the lesion or disease of the somatosensory nervous system OR a surgeon's clear verification of an intraoperative nerve lesion (intercostobrachial in MRM with Axillary Evacuation in Breast Surgery)
patient daily activity and functional capacity | 6 months after surgery
  Assessment of patient daily activity and functional capacity is evaluated using Eastern cooperative oncology group "ECOG" scoring, (0=fully active, 1= able to perform light effort, 2= in bed <50% of the day 3=in bed >50% of the day, 4=bed ridden, 5=died) so the low score the better.

SECONDARY OUTCOMES:
opioid consumption | Post-operative 24 hours
  opioid consumption using the Visual analogy scale (VAS) score,Post-operative opioid consumption measured by number of rescue dose of morphine 5mg IV administered when VAS was more than 4 and total requirement per 24 hours was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Salman, Principal Investigator — National Cancer Institute, Cairo Uneversity
Locations (1):
- National Cancer Institute Cairo University, Cairo, Egypt